CLINICAL TRIAL: NCT01258894
Title: Investigation of Human Alpha-fetoprotein Genes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jin-Chuan Sheu/ M.D. Ph.D., National Taiwan University Hospital
Other Study IDs: 201010019R
Record Dates: First submitted 2010-11-30; First posted 2010-12-13 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Elevated or Normal Alpha-fetoprotein Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 10c.c Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies revealed that patients with hereditary persistence of AFP also had persistent abnormal AFP. Therefore, this study will recruit the patients and their family with elevated AFP (>20 ng/mL) and normal AFP patients being control groups. Then, their AFP genes extracted from the blood will be analyzed.

DETAILED DESCRIPTION:
Abnormal AFP elevation was usually noted in liver regeneration, HCC, nonseminomatous germ cell tumors or other malignant tumors. However, some studies revealed that patients with hereditary persistence of AFP also had persistent abnormal AFP. Therefore, we study will recruit the patients and their family with elevated AFP (>20 ng/mL) and normal AFP patients being control groups. Then, their AFP genes extracted from the blood will be analyzed. The hypothesis of this study is that the mutation of AFP gene might be one of the causes of abnormal AFP.

ELIGIBILITY:
Inclusion Criteria:

* The patients and their family with elevated AFP (>20 ng/mL) and normal AFP patients being control groups. More than 20 years old

Exclusion Criteria:

* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients and their family with elevated AFP (>20 ng/mL) and normal AFP patients being control groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Chuan Sheu, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan